CLINICAL TRIAL: NCT01744561
Title: Effects of a Partially Supervised Conditioning Program in CF: an International Multi-centre, Randomized Controlled Trial
Brief Title: Effects of a Partially Supervised Conditioning Program in CF
Acronym: ACTIVATE-CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Prof. Helge Hebestreit, Professor Dr. med., Wuerzburg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT-CF-001
Record Dates: First submitted 2012-12-05; First posted 2012-12-06 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Cystic Fibrosis
Keywords: Exercise; Motivation; Feedback; web-based diary; pedometer
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental): Add three hours of intense physical activities per week to baseline activities. Weekly exercise should include at least 30 minutes of strength building activities and at least two hours of aerobic activities. Exercise bouts lasting 20 min or longer will be counted with respect to total weekly training time.
  Interventions: Behavioral: Exercise Intervention
- Control (No Intervention): Keep activity level constant

INTERVENTIONS:
Behavioral: Exercise Intervention — Add three hours of intense physical activities per week to baseline activities. Weekly exercise should include at least 30 minutes of strength building activities and at least two hours of aerobic activities. Exercise bouts lasting 20 min or longer will be counted with respect to total weekly training time.
  Arms: Exercise Intervention

SUMMARY:
Physical activity and exercise have become an accepted and valued component of Cystic Fibrosis care. Regular physical activity and exercise can slow the rate of decline of pulmonary function, improve physical fitness, and enhance quality of life. However, motivating people to be more active is challenging. Supervised exercise programs are expensive and labor intensive, and adherence falls off significantly once supervision ends. Unsupervised or partially supervised programs are less costly and more flexible, but compliance can be more problematic. The primary objective of this study is to evaluate the effects of a 12-months partially supervised exercise intervention along with regular motivation on forced expiratory volume in 1 second (FEV1) in a large international group of cystic fibrosis patients. Secondary endpoints include patient reported quality of life, as well as levels of anxiety and depression, and control of blood sugar. A total of 292 patients with cystic fibrosis 12 years and older with a FEV1 ≥35% predicted will be recruited. Following baseline assessments (2 visits) patients will be randomized into an intervention and a control group. Thereafter, they will be seen every 3 months for assessments in their centre for one year (4 follow-up visits). Along with individual counseling to increase vigorous physical activity by at least 3 hours per week on each clinic visit, the intervention group will document daily exercise and inactivity time and will receive a step counter and they will record their progress with a web-based program. They will also receive monthly phone calls from the study staff. After 6 months, they will continue with the step counter and web-based program for a further 6 months. The control group will receive access to this intervention after 12 months of standardized care. Should this relatively simple program prove successful, this will be made available on a wider scale internationally.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Cystic Fibrosis
* Age ≥12 years
* Forced expiratory volume in 1 second (FEV1) ≥ 35% predicted
* Access to the internet

Exclusion Criteria:

* Participation in another clinical trial up to 4 weeks prior to the first baseline visit
* Pregnancy/Breastfeeding
* Inability to exercise
* More than 4 hours of reported strenuous physical activities per week currently or up to 3 months prior to baseline measurements and not already planned within the coming 6 months.
* Unstable condition precluding exercise (major hemoptysis or pneumothorax within the last 3 months, acute exacerbation and iv-antibiotics during the last 4 weeks, planned surgery, listed for lung transplantation, major musculoskeletal injuries such as fractures or sprains during the last 2 months, others according to the impression of the doctor)
* Cardiac arrhythmias with exercise
* Requiring additional oxygen with exercise
* Recent diagnosis of diabetes 3 months prior to screening or at screening
* Recent changes in medication 1 month or less prior to screening (systemic steroids, ibuprofen, inhaled antibiotics, mannitol, DNAse, hypertonic saline)
* At least one G551D mutation and not on ivacaftor (VX770) yet but planned start or planned stop of ivacaftor during the trial
* Colonization with Burkholderia cenocepacia

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Change in forced expiratory volume in 1 second (FEV1; in % predicted using the average of two baseline measurements) from baseline to 6 months in the intervention group compared to controls. | baseline and 6 months

SECONDARY OUTCOMES:
Change in peak oxygen uptake (%predicted) | baseline to 6 months and baseline to 12 months
Change in maximal aerobic power (%predicted) | baseline to 6 months and baseline to 12 months
Change in measured steps per day | baseline to 6 months and baseline to 12 months
Change in exercise steps per day | baseline to 6 months and baseline to 12 months
Change in reported physical activity | baseline to 6 months and baseline to 12 months
Change in forced expiratory volume in 1 second (FEV1; %predicted) | baseline to 6 months and baseline to 12 months
Change in forced vital capacity (FVC; % predicted) | baseline to 6 months and baseline to 12 months
Change in residual volume in percent of total lung capacity (RV/TLC; %) | baseline to 6 months and baseline to 12 months
Time to first exacerbation | baseline to 6 months and baseline to 12 months
Number of upper respiratory tract infections | baseline to 6 months and baseline to 12 months
  from diary
Days on additional oral / intravenous antibiotics | baseline to 6 months and baseline to 12 months
  from questionnaire
Change in body mass index (kg/m2) | baseline to 6 months and baseline to 12 months
Change in muscle mass (kg) | baseline to 6 months and baseline to 12 months
  estimated from skinfold thickness
Change in percent body fat | baseline to 6 months and baseline to 12 months
  estimated from skinfold thickness
Change in Quality of Life scales | baseline to 6 months and baseline to 12 months
  from the revised Cystic Fibrosis health-related quality of life Questionnaire (CFQ-R questionnaire)
Change in depression, anxiety and stress scores | baseline to 6 months and baseline to 12 months
  from Depression Anxiety Stress Scales
Change in plasma glucose concentrations 1 and 2 hours after a standardized glucose load | baseline to 9 months
  standardized oral glucose tolerance test only patients without diabetes mellitus
Adverse events possibly or likely related to exercise | baseline to 6 months and baseline to 12 months
  causality as judged by investigator
Severe adverse events | baseline to 6 months and baseline to 12 months
Serious adverse events | baseline to 6 months and baseline to 12 months

OTHER OUTCOMES:
Compliance with the exercise goal | baseline to 6 months and baseline to 12 months
  based on questionnaire and diary
Change in lung clearance index | baseline to 6 months and baseline to 12 months
  based on nitrogen multiple breath washout, in selected centres only
Change in time spent in moderate-and-vigorous physical activity | baseline to 6 months and baseline to 12 months
  based on accelerometry, in selected centres only
Change in bone mineral density and body composition | baseline to 6 months and baseline to 12 months
  based on dual energy x-ray absorptiometry, in selected centres only
Change in mucociliary clearance with exercise | baseline to 6 months
  based on nuclear medicine scans, US centres only

CONTACTS AND LOCATIONS:
Overall Officials: Helge U Hebestreit, Dr. med., Principal Investigator — Wuerzburg University Hosptitals
Locations (28):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
- Austria (2):
  - Mukoviszidose-Ambulanz, Universitätsklinik für Kinder- und Jugendheilkunde,, Graz
  - Cystische Fibrose Zentrum für Kinder, Jugendliche und Erwachsene, Innsbruck
- Montreal Children's Hospital, McGill University Health Centre - Glen Site, Monrtreal, Quebec, Canada
- France (6):
  - Hôpital Renée Sabran, Service : Maladies respiratoires, Hyères
  - Hôpital Calmette, Service Pneumologie-immuno-allergologie boulevard du Pr Leclercq, Lille
  - Hôpital Jeanne de Flandre, Service: Pneumologie et allergologie pédiatriques, Lille
  - Hôpital Arnaud de Villeneuve, Service: Maladies respiratoires, Montpellier
  - Hôpital Necker, Service : Pneumologie et allergologie pédiatriques, Paris
  - Hôpital Maison Blanche, Service : Maladies respiratoires, Reims
- Germany (11):
  - Olgahospital, Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg
  - Klinik für Kinder- und Jugendmedizin, Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Children´s Hospital of the University, Würzburg, Bavaria
  - Pediatric Pulmonology and CF centre, Children´s Hospital, Ruhr University, Bochum
  - Klinik und Poliklinik für Kinderheilkunde - Universitäts-Mukoviszidose-Centrum, Dresden
  - Christiane Herzog CF-Zentrum, Goethe Universität, Frankfurt
  - CF Zentrum Hamburg-Altona, Kinderarztpraxis Runge, Sextro,Held, Hamburg
  - CF- Ambulanz, Kinderklinik, Pädiatrische Pneumologie, Allergologie und Neonatologie, Hanover
  - Zentrum für Kinder- und Jugendmedizin, Pädiatrische Pneumologie, Allergologie und Mukoviszidose, Mainz
  - Praxis für Lungen- und Bronchialheilkunde, Munich
  - Klinik für Kinder- und Jugendmedizin / Universitätsklinikum, Münster
- University Medical Center, Child Development & Exercise Center, Wilhelmina Children's Hospital, Utrecht, Netherlands
- Switzerland (4):
  - QuartierBleu, Praxis für Pneumologie am Lindenhofspital, Bern
  - Inselspital, Universitätsklinik für Kinderheilkunde, Pneumologie, Bern
  - Kinderspital, Pneumologie, Zurich
  - UniversitätsSpital, Klinik für Pneumologie, Zurich
- Royal Hospital for Sick Children, Edinburgh, Scottland, United Kingdom

REFERENCES:
- [Background] Hebestreit H, Lands LC, Alarie N, Schaeff J, Karila C, Orenstein DM, Urquhart DS, Hulzebos EHJ, Stein L, Schindler C, Kriemler S, Radtke T; ACTIVATE-CF Study Working Group. Effects of a partially supervised conditioning programme in cystic fibrosis: an international multi-centre randomised controlled trial (ACTIVATE-CF): study protocol. BMC Pulm Med. 2018 Feb 8;18(1):31. doi: 10.1186/s12890-018-0596-6. PMID 29422091